CLINICAL TRIAL: NCT05910112
Title: Prospective Data Collection on Clinical, Radiological and Patient Reported Outcomes After Pleural Intervention
Acronym: PROSPECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Beckton Dickinson (Unknown)
Responsible Party: Sponsor
Other Study IDs: 260269
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pleural Diseases; Pleural Mesothelioma; Pneumothorax; Pleural Effusion; Pleural Infection; Pleural Neoplasms; Pleural Metastases; Pleural Effusion, Malignant; Procedural Complication; Complications, Pulmonary
MeSH Terms: conditions — Pleural Diseases; Mesothelioma, Malignant; Pneumothorax; Pleural Effusion; Pleural Neoplasms; Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undergoing pleural intervention: Any patient undergoing a pleural procedure (eg thoracocentesis, chest drain, indwelling pleural catheter, pleural biopsies, medical thoracoscopy)
  Interventions: Procedure: Pleural interventions

INTERVENTIONS:
Procedure: Pleural interventions — eg thoracocentesis, chest drain, indwelling pleural catheters, thoracoscopy

SUMMARY:
The PROSPECT study aims to look at the number of problems or side effects which occur after patients have had a procedure completed to remove fluid or air from the space between the lung and the chest wall. Other information will also be collected to see whether anything else affects which patients have problems after the procedure such as bleeding or infection. This study will also investigate whether it is possible to find out which patients are likely to feel a lot better after the procedure. Not all patients feel significantly better but it is not clear why this is. There are a number of different reasons patients may not feel better, for example if the lung is not able to fully re-expand. The study aims to look at whether it is possible to predict these problems before the procedure using ultrasound. If it is possible to find the answers to some of these questions it might be possible to prevent patients undergoing treatments which are not likely to benefit them. The study will use information already collected as part of clinical care, as well as questionnaires from patients receiving care at a variety of centres. The different features of these centres will also be considered in analysis.

DETAILED DESCRIPTION:
PROSPECT is a prospective, observational study in which complications and key other data will be collected from patients undergoing pleural procedures. Data will include demographics, smoking history, pre-procedure observations, radiological findings and medical history along with information about the size of the service and range of procedures performed. Complications will be objectively defined, with baseline procedure information recorded, and at 1 month, all complications recorded according to specified criteria.

At least 20 centres will be approached to collect prospective data on pleural interventions and outcomes for patients who have undergone procedures in their service. All patients who have a pleural procedure for fluid will have an ultrasound as part of the procedure but due to a difference in expertise around the country, centres (and clinicians within each centre) will record ultrasound findings in varying degrees of detail. Centres will specify what level of detail they can provide and can opt to perform a more detailed assessment if skills permit and the patient agrees. Any patient can be included in the sub-study if there is sufficient time and sufficient expertise of the clinicians to perform and interpret the more detail scanning procedures.

Patients, who are willing, will also be asked to complete a visual analogue scale score for chest pain and breathlessness before and after their procedure and at a further time interval within 4 weeks. Any patients who are having an indwelling catheter inserted, or chest drain inserted for pleurodesis will be asked to complete an additional questionnaire.

The majority of centres will be those with an active pleural service and will include a combination of district general and tertiary referral centres. The data is likely to represent best practice but should also include the complex cases and interventions. In the future, the study is extendable to non-specialist centres to achieve similar reporting standards, mirroring current standards in other areas such as surgery. The data collected will provide a "best practice standard" against which new and smaller volume centres can benchmark practice, to ensure patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18
* Undergoing pleural intervention
* Able to provide written informed consent

Exclusion Criteria:

* Aged <18
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Patients undergoing invasive pleural intervention in a variety of settings: day case procedure lists, pleural clinic, bedside
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Complications | within 30 days
  Specifically: bleeding, infection, pneumothorax, organ injury, pain, re-expansion pulmonary oedema

SECONDARY OUTCOMES:
Patient reported outcome measures of dyspnoea and chest pain | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Najib Rahman, DPhil, Study Chair — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided